CLINICAL TRIAL: NCT03029598
Title: Anti-PD-1 Therapy in Combination With Platinum Chemotherapy for Platinum Resistant Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Brief Title: Pembrolizumab and Carboplatin in Treating Patients With Relapsed or Refractory Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, John Liao, Associate Professor, Division of Gynecologic Oncology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9740; NCI-2016-01962 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9740 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1716074 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Results first posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Carboplatin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, carboplatin) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and carboplatin IV over 30 minutes on days 8 and 15. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase I/II trial studies how well pembrolizumab and carboplatin work in treating patients with ovarian, fallopian tube, or primary peritoneal cancer that has come back (relapsed) or has not responded to previous treatment (refractory). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pembrolizumab and carboplatin with platinum resistant chemotherapy may work better than platinum chemotherapy alone in treating patients with ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the clinical response rate of platinum chemotherapy and pembrolizumab (MK-3475) in platinum chemotherapy pretreated ovarian, fallopian tube, and primary peritoneal.

II. To examine whether retreatment with platinum chemotherapy in platinum resistant ovarian, fallopian tube, and primary peritoneal cancers improves progression free survival by concurrent administration of MK-3475.

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of concurrent administration of MK-3475 with platinum chemotherapy in patients with platinum resistant recurrent ovarian, fallopian tube, and primary peritoneal cancers.

II. To determine the relationship between PD-L1 expression and response to the combination of MK-3475 and platinum.

III. To assess the overall survival of patients treated with the combination of MK-3475 and platinum.

EXPLORATORY OBJECTIVE:

I. To explore whether treatment with MK-3475 and platinum alters soluble factors in sera, peripheral immune responses and immune cell profile.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and carboplatin IV over 30 minutes on days 8 and 15. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year, every 6 months for 1 year, and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of ovarian, fallopian tube, or primary peritoneal cancer patients who had a complete response to primary treatment with platinum based chemotherapy, have progressed within 6 months of completing platinum based chemotherapy and have subsequently received at least one, non-platinum-based, therapy
* Have relapsed, refractory, or progressive disease following last line of treatment
* Have estimated life expectancy of at least 3 months
* Be willing and able to provide written informed consent/assent for the trial
* Have measurable disease with at least 1 unidimensional lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500/mcL (within 10 days of treatment initiation)
* Platelets >= 100,000/mcL (within 10 days of treatment initiation)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment) (within 10 days of treatment initiation)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (within 10 days of treatment initiation)

  *Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (within 10 days of treatment initiation)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases (within 10 days of treatment initiation)
* Albumin >= 2.5 mg/dL (within 10 days of treatment initiation)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 10 days of treatment initiation)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (within 10 days of treatment initiation)
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment

  * Short-term administration of systemic steroids (i.e., for allergic reactions or the management of immune related adverse events [irAEs]) is allowed
* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Clinically significant cardiovascular disease
* Known severe hypersensitivity reactions to monoclonal antibodies or carboplatin >= grade 3, any history of anaphylaxis, or uncontrolled asthma
* Has received prior therapy with pembrolizumab
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Liao, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Liao JB, Gwin WR, Urban RR, Hitchcock-Bernhardt KM, Coveler AL, Higgins DM, Childs JS, Shakalia HN, Swensen RE, Stanton SE, Tinker AV, Wahl TA, Ancheta RG, McGonigle KF, Dai JY, Disis ML, Goff BA. Pembrolizumab with low-dose carboplatin for recurrent platinum-resistant ovarian, fallopian tube, and primary peritoneal cancer: survival and immune correlates. J Immunother Cancer. 2021 Sep;9(9):e003122. doi: 10.1136/jitc-2021-003122. PMID 34531249

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, Carboplatin)
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, Carboplatin)
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 65 [41 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28
  Canada | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR) Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI/CT scans: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Carboplatin)
Number analyzed (Participants) | 23
Participants
  Patients that achieved a Partial Response (PR) | 3
  Patient achieved Stable Disease (SD) | 15
  Patients that had Progressive Disease (PD) | 5

2. Primary Outcome: Progression-free Survival (PFS) Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Analyzed using the Kaplan-Meier method. Kaplan-Meier estimates of the survival function with 95% confidence intervals (CIs) at specific time points (using Greenwood's formula for the standard error) were computed. Comparisons with the historical control PFS will be conducted by examining whether the 95% confidence internal covers the historical control proportions.
  Progression-free survival (PFS) is defined as the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse. Participants are evaluated by RECIST1.1 to determine if/when a participant's disease has progressed defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Carboplatin)
Number analyzed (Participants) | 29
months | 4.63 [4.30 to 4.97]

3. Secondary Outcome: Count of Adverse Events Evaluated by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Description: The safety evaluation of the population included all patients who received at least one dose of study medication. The descriptions and grading scales found in the revised NCI CTCAE version 4.0 will be utilized for adverse event reporting where Grade refers to the severity of the AE.
  The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:
  Grade 1 Mild; asymptomatic or mild symptoms Grade 2 Moderate; minimal Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care of activity of daily living Grade 4 Life-threatening consequences; urgent intervention indicated Grade 5 Death related to AE
Time Frame: Up to 3.5 years
Measure: Number; unit: adverse events
Arm/Group | Treatment (Pembrolizumab, Carboplatin)
Number analyzed (Participants) | 29
adverse events
  Grade 1 - Total Number of Reported AEs | 597
  Grade 2 - Total Number of Reported AEs | 169
  Grade 3 - Total Number of Reported AEs | 40
  Grade 4 - Total Number of Reported AEs | 2

4. Secondary Outcome: Number of Participants That Were PD-L1 Positive Based On PD-L1 Expression of Primary Tumor Blocks Assessed by Immunohistochemical Staining
Description: PD-L1 antibody-stained archival tumor was evaluated by a board-certified pathologist and given a modified proportion score (MPS), or the overall percent of positive cells expressing PD-L1, and a MPS ≥ 5% was defined as PD-L1 positive.
Time Frame: Up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Carboplatin)
Number analyzed (Participants) | 23
Participants | 7

5. Secondary Outcome: Overall Survival (OS)
Description: Analyzed using the Kaplan-Meier method. Kaplan-Meier estimates of the survival function with 95% CIs at specific time points (using Greenwood's formula for the standard error) were computed. Comparisons with the historical control OS will be conducted by examining whether the 95% confidence internal covers the historical control proportions.
Time Frame: Up to 3.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Carboplatin)
Number analyzed (Participants) | 29
months | 11.3 [6.094 to 16.506]

6. Secondary Outcome: Best Overall Response (BOR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI/CT scans: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Carboplatin)
Number analyzed (Participants) | 23
Participants
  Partial Response | 3
  Stable Disease | 15
  Progressive Disease | 5

7. Secondary Outcome: Progression-free Survival (PFS) Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Analyzed using the Kaplan-Meier method. Kaplan-Meier estimates of the survival function with 95% CIs at specific time points (using Greenwood's formula for the standard error) were computed. Comparisons with the historical control PFS will be conducted by examining whether the 95% confidence internal covers the historical control proportions.
  Progression-free survival (PFS) is defined as the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse. Participants are evaluated by RECIST1.1 to determine if/when a participant's disease has progressed defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 3.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Carboplatin)
Number analyzed (Participants) | 29
months | 4.63 [4.3 to 4.97]

8. Secondary Outcome: Immune-related Best Overall Response (BOR) Assessed Using irRECIST (Immune-related Response Evaluation Criteria In Solid Tumors) Derived From Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: as for outcome 1
Time Frame: Up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Carboplatin)
Number analyzed (Participants) | 23
Participants
  Partial Response | 3
  Stable Disease | 15
  Progressive Disease | 5

9. Secondary Outcome: Immune-related Progression-free Survival (PFS) Using irRECIST (Immune-related Response Evaluation Criteria In Solid Tumors) Derived From Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Progression-free survival (PFS) is defined as the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse. Participants are evaluated by RECIST1.1 to determine if/when a participant's disease has progressed defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 3.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Carboplatin)
Number analyzed (Participants) | 29
months | 4.63 [4.30 to 4.97]

ADVERSE EVENTS:
Time Frame: The safety population included all patients who received at least one dose of study medication. Anyone that received at least 1 treatment dose will be evaluated. After the end of treatment, each subject will be followed for 30 days or prior to initiation of new treatment for adverse event monitoring (serious adverse events will be collected for 90 days after the end of treatment. The complete adverse event evaluation period for all treated participants is 3.5 years.
Description: We used CTCAE v4.0 for this study. The adverse events reported here include all events regardless of whether they were unrelated and related to study treatment). Please note we recorded every adverse event for every subject regardless of severity. For example, a subject may have an injection site reaction at the site of treatment administration; each each time an injection site reactions is reported, during the study, it is recorded for that subject.
Arm/Group | Treatment (Pembrolizumab, Carboplatin)
All-Cause Mortality (participants affected / at risk) | 28/29
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 25/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Carboplatin) (N=29)
Disease progression leading to hospice (General disorders) | 1 (1) — For this study disease progression was not defined as an SAE, unless it led to hospitalization or death
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Carboplatin) (N=29)
Lymphopenia (Investigations) | 19 (100) — 3 reported adverse events were deemed unrelated to study treatment
Anemia (Blood and lymphatic system disorders) | 25 (82) — 31 reported adverse events were deemed unrelated to study treatment
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 (42) — 18 reported adverse events were deemed unrelated to study treatment
Thrombocytopenia (Investigations) | 13 (37) — 4 reported adverse events were deemed unrelated to study treatment
White blood cell decreased (Investigations) | 14 (35) — 2 reported adverse events were deemed unrelated to study treatment
Hypocalcemia (Metabolism and nutrition disorders) | 14 (31) — 24 reported adverse events were deemed unrelated to study treatment
Hypokalemia (Metabolism and nutrition disorders) | 14 (27) — 23 reported adverse events were deemed unrelated to study treatment
Nausea (Gastrointestinal disorders) | 13 (26) — 5 reported adverse events were deemed unrelated to study treatment
Neutropenia (Investigations) | 7 (25)
Hypomagnesemia (Metabolism and nutrition disorders) | 14 (24) — 6 reported adverse events were deemed unrelated to study treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT03029598/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT03029598/ICF_001.pdf